CLINICAL TRIAL: NCT06127472
Title: Support With Psychoeducation for Older Adults With Autism Study
Brief Title: Psychoeducation for Older Adults With Autism
Acronym: OPAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Collaborators: GGZ Breburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL84067.028.23
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; older adults
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: The effects of the adapted PE program will be evaluated in a Stepped Wedge Trial Design (SWTD), with the intervention sequentially rolled-out in eleven (specialised) mental healthcare organisations. Furthermore, a pre-post design will be used to compare the situation before the roll-out period with the situation after the roll-out period.
  A second intervention, training and education in detection and diagnosis of ASD in older adults, is rolled out in de same SWTD. The effects of this intervention will also be assessed further in pre-post design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ASD trained (Other): Periods in the SWTD after receiving training in detection and diagnosis of ASD.
  Interventions: Other: Training in detection and diagnosis of ASD
- ASD training - control (Other): Periods in the SWTD before receiving training in detection and diagnosis of ASD.
  Interventions: Other: Training in detection and diagnosis of ASD
- PE program (Other): Periods in the SWTD after receiving the PE program.
  Interventions: Other: PE program
- PE program - control (Other): Periods in the SWTD before receiving the PE program.
  Interventions: Other: PE program

INTERVENTIONS:
Other: Training in detection and diagnosis of ASD — To improve detection and diagnosis of ASD the participating mental health institutes will be trained by the research group on how to detect and diagnose autism in older adults. The basis of the ASD training involves two separate training sessions. Part one focuses on recognition and detection of ASD, specifically in older adults, and will be offered to the entire teams of the participating centres. The second part of the training focuses on the diagnosis of ASD and as such is offered primarily to diagnosticians. Follow up will consist of monthly recurring options for online consultation during the entire project to discuss clinical cases by experts in ASD in older adults from PersonaCura, clinical centre of excellence for personality and developmental disorders in older adults (dr. A. Videler and R. Wilting).
  Arms: ASD trained; ASD training - control
Other: PE program — An adapted PE program for older adults with a (probability) diagnosis of ASD. The PE program consists of eight, two-hour group meetings on a weekly basis.
  Arms: PE program; PE program - control

SUMMARY:
Until recently, autism in older adults went unrecognised. Although there has been more attention to autism in older adults in recent years, there is still a lot of unfamiliarity with the phenomenon and underdiagnosis in (mental) health care. Many care providers are reluctant to diagnose autism in later life, due to a lack of knowledge about autism in older adults and because there is still very little scientific knowledge available for this target group. Although several multidisciplinary guidelines for autism in adults prescribe that after the diagnosis psycho-education is the first step in treatment, psycho-education is still only offered in a few places in the Netherlands. Psycho-education is important to help older people gain knowledge about their autism, to help them understand and accept this diagnosis, in order to subsequently make the treatment of the problems, with which they turn to the mental health care, more appropriate and effective.

The aim of this study is to contribute to better recognition and diagnosis of autism among older adults. This research also aims to improve a psycho-education program for older adults and investigate its effects.

The scientific research question is whether training in ASD for health care professionals results in better recognition and detection of ASD in older adults, and whether participation in the psycho-education course for older adults, who have been diagnosed with autism, or have received a probability diagnosis ASD, contributes to improvement of mental health and quality of life.

DETAILED DESCRIPTION:
The detection of autism spectrum disorder (ASD) in older adults in Dutch (specialised) mental health care is improving, but underdiagnosis remains. Older adults with ASD experience a low quality of life (QoL) and a high rate of psychopathology across the life span and into old age. Additionally, Dutch and international treatment guidelines advocate psychoeducation (PE) as the first intervention after patients have been diagnosed with ASD. However, as PE for older patients with ASD is hardly available in the Netherlands, access to PE is severely limited for these older adults. Hence, it is important to improve detection and diagnosis of ASD and increase the availability of PE for older adults. The hypotheses of this study are 1) that detection and diagnosis of ASD in older adults will significantly increase following training of professionals and 2) that delivering an adapted and improved PE program for older adults will result in more knowledge and recognition of ASD, a better acceptance of the diagnosis, improved coping with ASD, improved resilience and comorbid general psychological distress, and ultimately in higher quality of life, compared to those patients with ASD that receive no PE.

The aim of this study on the one hand is to gain insight into: 1) the effects of providing training and education to mental health care providers in detection and diagnosis of ASD in older adults, with the expectation that this contributes to an increase in the number and proportion of ASD diagnoses in older adults in the Netherlands; 2) the effects of a PE program for older adults with ASD in terms of knowledge and recognition of ASD and traits, a better acceptance of the diagnosis, improved coping with ASD, improved resilience and comorbid general psychological distress - and ultimately higher quality of life; and 3) the experiences of older adults with ASD following the PE program.

Study design: The effects of training and education in detection and diagnosis of ASD in older adults, and the effects of the PE program will be evaluated in a Stepped Wedge Trial Design (SWTD), with the intervention sequentially rolled-out in eleven (specialised) mental healthcare organisations. Furthermore, a pre-post design will be used to compare the situation before the roll-out period with the situation after the roll-out period in terms of diagnosis and individual outcomes such as knowledge regarding ASD. Qualitative measures will be used to assess the experiences of older adults with ASD who participated in the PE program.

Study population: Older adults - aged 55 and over diagnosed with ASD or a probability diagnosis by a multidisciplinary team according to the Dutch multidisciplinary guidelines, as confirmed by the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) interview for ASD, or the Netherlands Interview for Diagnosis of ASD in adults (NIDA) as well as a proxy (an individual who provides reports on behalf of, or about, a study participant).

The intervention consists of education in detection and diagnosis of ASD in older adults for mental health professionals and of an adapted PE program for older adults with a (probability) diagnosis of ASD. The PE program consists of eight, two hour group meetings on a weekly basis.

Primary study parameter concerns clinical outcomes measuring effects of the psycho-education course in terms of quality of life, acceptance of the diagnosis, knowledge of ASD, recognition of ASD traits, coping with ASD, quantitative autistic traits, resilience, and comorbid psychological distress. Quality of life is assessed by the MHQoL-7 (Mental Health Quality of Life Questionnaire). Acceptance of the diagnosis, knowledge and coping with ASD are assessed with use of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis (VKHAA). Acceptance of ASD (-diagnosis) is further assessed through the Acceptance Questionnaire (AQ). Autistic traits are assessed through the Social Responsiveness Scale-Adults (SRS-A). Comorbid psychological distress is assessed by the Brief Symptom Inventory (BSI). All these assessments are performed (1) at baseline (following diagnosis and informed consent); (2) before the patient starts with PE (on average three months after baseline; participants in the control group will receive this three months after baseline; (3) after the PE (on average two months after the start of the PE program; participants in the control group will receive this measurement 6 months after baseline); (4) at 9-months follow-up (nine months after second measurement). A proxy, chosen by the study participant, will additionally inform on acceptance, knowledge, recognition, coping and ASD traits through measurements on the VKHAA for informants (VKHAA-N) and SRS-A for informants (SRS-A-N) at two moments that overlap with measurements 2 and 3 of study participants.

Secondary study parameters is the number and proportion of ASD diagnoses in the participating centres (collected from the information and registration systems of the mental health care centres) from one year before, during the project, and at one year follow-up.

For patients, benefits will be considerable as they will receive a PE program that is recommended by the Dutch multidisciplinary guideline for ASD in adults, and although being the recommended first intervention by treatment guidelines, is not provided to them momentarily. The benefits account for patients who provide informed consent to participate in the research and patients who do not give their consent, since the same treatment will be available for both. The investigators consider the burden of participating in the research, which consists of filling out questionnaires and inviting a proxy of their choice to fill out two of the same questionnaires, to be limited. Firstly, because this will be done in the context of treatment that fits the recommended first intervention by treatment guidelines and thus does not provide an extra mental burden. Moreover, the time needed to fill out these questionnaires is limited: approximately 40 to 60 minutes per measurement point, and there are no indications that risks are involved with regard to the topics of these questionnaires; specifically in a similar study by the study's research group, no adverse events or risks were observed.

Additional potential benefits exist in the form of increased detection and diagnosis of ASD in older adults across participating organisations, while the burden of participating in the study hardly exceeds time and effort spent in diagnostic efforts as usual, yet lightens efforts spent on informing patients with an ASD diagnosis as this can be done in a group format rather than on an individual basis. The only extra effort is limited to informing patients about the study with verbal and written information.

ELIGIBILITY:
Inclusion Criteria:

* minimum of 55 years old.
* diagnosed with ASD or a probability diagnosis by a multidisciplinary team according to the Dutch multidisciplinary guideline, as confirmed by the DSM-5 interview for ASD (Spek, n.d.), or the Netherlands Interview for Diagnosis of ASD in adults (NIDA; Vuijk, 2023)

Exclusion Criteria:

* comorbid mental disorder that needs acute treatment and severely interferes with a group treatment (for example psychosis),
* a major neurocognitive disorder (for example dementia or acquired brain injury),
* substance abuse disorder, that requires detoxification, and/or
* an IQ below 70.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life (MHQoL-7) | minimum of 9 to maximum of 15 months with four measurements over this period.
  Quality of life as measured with the Mental Health Quality of Life-7 (MHQoL-7) a standardized quality of life questionnaire specifically aimed at people with mental health problems. The MHQoL-7D index score can vary from 0 to 21, with higher scores indicating better quality of life.
Acceptance of the diagnosis | minimum of 9 to maximum of 15 months with four measurements over this period.
  Acceptance of the diagnosis is based on the combined scores from patients and their chosen proxy on item 31 of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis (VKHAA and VKHAA-N for proxies). The score on this item is binary with either yes or no scores. Scores thus range from 0 to 1, with a score of 1 reflecting acceptance as opposed to a score of 0 (no acceptance). This data further is aggregated with measurements of patients' acceptance of the diagnosis as evaluated with the Acceptance Questionnaire (AQ), a questionnaire with scores ranging from 0 to 33 and higher scores reflecting higher diagnosis acceptance. Total acceptance scores thus have a range from 0 - 35 and higher scores indicating more acceptance.
Acceptance of the diagnosis from proxy perspective | 8 weeks with two measurements over this period.
  Acceptance of the diagnosis as reflected by proxies is based on item 31 from the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis for Proxies (VKHAA-N). The score on this item is binary with either yes or no scores. Scores thus range from 0 to 1, with a score of 1 reflecting acceptance as opposed to a score of 0 (no acceptance).
Knowledge of ASD | minimum of 9 to maximum of 15 months with four measurements over this period.
  Knowledge of ASD is based on measurements on items 1-18 of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis (VKHAA). Scores range from 0 to 54 with higher scores indicating more knowledge of ASD.
Knowledge of ASD from proxy perspective | 8 weeks with two measurements over this period.
  Knowledge of ASD as reflected by proxy perspective is based on measurements on items 1-18 of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis for Proxies (VKHAA-). Scores range from 0 to 54 with higher scores indicating more knowledge of ASD.
Recognition of ASD traits | minimum of 9 to maximum of 15 months with four measurements over this period.
  Recognition of ASD is based on measurements on items 20-25 of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis (VKHAA). Minimum to maximum values are 0 through 24, with higher scores reflecting more recognition of ASD.
Recognition of ASD traits from proxy perspective | 8 weeks with two measurements over this period.
  Recognition of ASD as reflected by the proxy perspective is based on measurements on items 20-25 of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis for Proxies (VKHAA-N). Minimum to maximum values are 0 through 24, with higher scores reflecting more recognition of ASD.
Coping with ASD | minimum of 9 to maximum of 15 months with four measurements over this period.
  Coping with ASD is based on measurements on items 19 and 28-30 of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis (VKHAA). Scores range from 0 to 15, with higher scores indicating better coping with ASD.
Coping with ASD from proxy perspective | 8 weeks with two measurements over this period.
  Coping with ASD from the proxy perspective is based on measurements on items 19 and 28-30 of the Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis for Proxies (VKHAA-N). Scores range from 0 to 15, with higher scores indicating better coping with ASD.
Quantitative autistic traits | minimum of 9 to maximum of 15 months with four measurements over this period.
  Autistic traits are evaluated with use of the Social Responsiveness Scale-Adults (SRS-A). The questionnaire consists of 4 subscales: Social Awareness (SA), Social Communication (SC), Social Motivation (SM) and Repetitiveness and Rigidity (RR). Scores on the SRS-A range from 64 to 256 with higher scores reflecting more autistic traits.
Quantitative autistic traits from proxy perspective | 8 weeks with two measurements over this period.
  Autistic traits from the proxy perspective are evaluated with use of the Social Responsiveness Scale-Adults for proxies, the SRS-A-N. The questionnaire consists of 4 subscales: Social Awareness (SA), Social Communication (SC), Social Motivation (SM) and Repetitiveness and Rigidity (RR). Scores on the SRS-A-N range from 64 to 256 with higher scores reflecting more autistic traits.
Resilience | minimum of 9 to maximum of 15 months with four measurements over this period.
  Resilience will be assessed with a 10-item questionnaire, the Connor-Davidson Resilience Scale (CD-RISC-10). Scores range from 0 - 40 with higher scores indicating greater resilience.
Comorbid psychological distress | minimum of 9 to maximum of 15 months with four measurements over this period.
  Comorbid psychological distress will be assessed through the Brief Symptom Inventory (BSI). BSI is a 53-item questionnaire with 9 subscales for somatic complaints, cognitive problems, interpersonal sensitivity, depressive mood, anxiety, hostility, phobia, paranoia and psychoticism. Scores range from 0 - 212 with higher scores indicating higher presence of psychological complaints.

SECONDARY OUTCOMES:
Number of ASD diagnoses | Collection of data concerns numbers per month, starting from one year before, during the expected 18 months of the roll out of the ASD training intervention, and at one year follow-up following roll out of this training in the last cluster of the SWTD.
  The number of ASD diagnoses collected from the information and registration systems of the participating mental health care centres.
Proportion of ASD diagnoses | Collection of data concerns numbers per month, starting from one year before, during the expected 18 months of the roll out of the ASD training intervention, and at one year follow-up following roll out of this training in the last cluster of the SWTD.
  The proportion of ASD diagnoses collected from the information and registration systems of the participating mental health care centres.

OTHER OUTCOMES:
Descriptives | At informed consent (zip code) and the baseline measurement (gender, age, education level), which averages the first two weeks of participants' inclusion in the study.
  For descriptives, demographic information, concerning gender, age, zip code and education level will be gathered.

CONTACTS AND LOCATIONS:
Overall Officials: Arjan Videler, Dr., Principal Investigator — Tilburg University, GGz Breburg
Locations (11):
- Netherlands (11):
  - GGNet Ouderen (Elderly), Apeldoorn, Gelderland
  - Mondriaan Ouderen (Elderly), Heerlen, Limburg
  - Vincent van Gogh Ouderen (Elderly), Venray, Limburg
  - Reinier van Arkel, 's-Hertogenbosch, North Brabant
  - GGzE Nestor, Eindhoven, North Brabant
  - SeneVita GGZ, Eindhoven, North Brabant
  - GGz WNB Ouderen (Elderly), Halsteren, North Brabant
  - GGz Breburg PersonaCura, Tilburg, North Brabant
  - GGz NHN Frailty, Hoorn, North Holland
  - GGz Mediant, Enschede, Overijssel
  - Dimence, Deventer

IPD SHARING:
Plan to Share IPD: No
Data will be saved on the secured server of Tranzo, Tilburg University, for 15 years. Three years after the research project is completed, other researchers may apply to use the research data. This concerns only processed and fully anonymized data. Only applications for research that has a purpose similar to the purpose of the current study may be approved. Participants that do not want their data used for this purpose can indicate so on their consent form. They will still be able to participate in the study and will receive the same treatment in that case.

REFERENCES:
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] de Beurs, E. (2011). Brief Symptom Inventory-BSI. Handleiding herziene editie 2011. Leiden: PITS BV.
- [Background] Cage E, Di Monaco J, Newell V. Experiences of Autism Acceptance and Mental Health in Autistic Adults. J Autism Dev Disord. 2018 Feb;48(2):473-484. doi: 10.1007/s10803-017-3342-7. PMID 29071566
- [Background] van Krugten FCW, Busschbach JJV, Versteegh MM, Hakkaart-van Roijen L, Brouwer WBF. The Mental Health Quality of Life Questionnaire (MHQoL): development and first psychometric evaluation of a new measure to assess quality of life in people with mental health problems. Qual Life Res. 2022 Feb;31(2):633-643. doi: 10.1007/s11136-021-02935-w. Epub 2021 Jul 9. PMID 34241821
- [Background] Verbeek, I.C., Wedjelek, J., Elfeddali, I., & Videler, A.C. (2023). Acceptance Questionnaire Dutch translation. In development.
- [Background] Verbeek, I.C., Lenders, M.A.C.., van Alphen, S.P.J., Elfeddali, I., & Videler, A.C., (2023a). Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis. In development.
- [Background] Verbeek, I.C., Lenders, M.A.C, van Alphen, S.P.J., Elfeddali, I., & Videler, A.C., (2023b). Questionnaire Knowledge, Recognition and Acceptance of Autism Diagnosis for Proxies. In development.
- [Background] Constantino, J.N., & Gruber, C.P. (2016). SRS-A Screeningslijst voor autismespectrumstoornissen: Handleiding. Hogrefe. [Dutch Handbook for the Social Responsiveness Scale for Adults]